CLINICAL TRIAL: NCT05529537
Title: The Effect of Manual Lymphatic Drainage on Upper Extremity Functionality in Rheumatoid Arthritis Patients
Brief Title: Manual Lymphatic Drainage for Rheumatoid Arthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Selcuk University (Other)
Responsible Party: Principal Investigator, Emine Cihan, principal investigator, Selcuk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022/08-01
Record Dates: First submitted 2022-09-01; First posted 2022-09-07 (Actual); Last update posted 2022-12-19 (Actual); Status verified 2022-12

CONDITIONS: Effect of Manual Lymphatic Drainage on Upper Extremity Functionality in Rheumatoid Arthritis
MeSH Terms: interventions — Manual Lymphatic Drainage

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control (Active Comparator)
  Interventions: Other: excersize
- MLD (Experimental)
  Interventions: Other: manual lymphatic drainage; Other: excersize

INTERVENTIONS:
Other: manual lymphatic drainage — In addition to conventional treatment for 4 weeks, manual lymph drainage will be applied to the patients.
  Arms: MLD
Other: excersize — upper extremity normal joint range of motion exercise, strengthening exercise, tendon gliding exercises

SUMMARY:
Rheumatoid arthritis (RA) is a chronic, progressive, autoimmune disease characterized by inflammation of the synovial joints and tendon sheaths. As a result of synovitis, progressive damage occurs in cartilage, bone and joints. This damage leads to severe functional limitations and deterioration in quality of life. Synovial tissues are the main site of involvement. Manual lymph drainage reduces the levels of inflammatory mediators associated with edema and pain in the acute phase. On the basis of this concept; Stimulating the lymph system and increasing circulation, removing biochemical residues, regulating sympathetic and parasympathetic system responses, and thus reducing edema and pain. The increase in cardiac parasympathetic activity measured after MLD also contributes to relaxation. In addition to the transport of lymphatic fluid, manual lymph drainage stimulates free nerve endings in the skin with the touches it contains. Gentle stimulation to the skin increases tactile input and closes the pain pathways. In addition, the superficial relaxation and warming provided by soft stimulation creates an effect on the autonomic nervous system and activates the parasympathetic system. The aim of this study is to evaluate the effect of manual lymphatic drainage on upper extremity functionality in individuals with rheumatoid arthritis.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with RA according to ACR criteria
* Being between the ages of 18-65
* Volunteering to participate in the study

Exclusion Criteria:

* Presence of neuromuscular disease
* Having difficulty walking
* Cognitive impairment
* Having systemic disease such as diabetes mellitus and osteoarthritis
* History of upper extremity sIf you have Hand Deformity

Ages: 25 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2022-08-17 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-10-01 (Actual)

PRIMARY OUTCOMES:
Rheumatoid Arthritis Quality of Life Scale (QOL-RA) | 10 minutes
  In the scale consisting of 30 questions; questions are scored as "yes-1" and "no-0". The scores obtained range from 0-30, and high scores indicate poor quality of life.
pressure pain threshold | 5 minutes
  It is used for the assessment of sensitivity to pain and the determination of pressure perception. will be evaluated with a digital algometer device with a surface area of 1 cm2 and a sensitivity of 0.25 kg/cm2 (Jtech Medical Industries, ZEVEX Company, USA).
hand grip strength | 5 minutes
  The Jamar hand dynamometer, which is recommended by the American Association of Hand Therapists (AETD) and has high validity and reliability in many studies and is therefore accepted as the gold standard, will be used.
finger grip strength | 5 minutes
  Finger pinchmeter (Baseline) will be used to measure finger grip strength.

CONTACTS AND LOCATIONS:
Locations (1):
- Kutahya Health Science University Hospital, Kütahya, Turkey (Türkiye)